CLINICAL TRIAL: NCT04817514
Title: "Shoulder Musculoskeletal Disorders in Type 2 Diabetes Mellitus: Contributing Factors and Rehabilitation Protocol"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Católica del Maule (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Fernanda Assis Paes Habechian, Principal investigator, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11200574
Record Dates: First submitted 2021-03-16; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 2; Musculoskeletal Pain; Shoulder Pain
Keywords: Diabetes mellitus; Shoulder function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Musculoskeletal Pain; Shoulder Pain; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to what kind of protocol the participant is going through
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- specific shoulder rehabilitation protocol group (SRG); (Experimental)
  Interventions: Other: Shoulder rehabilitation exercises and aerobic exercises
- specific protocol of shoulder rehabilitation plus aerobic exercise group (ARG) (Experimental)
  Interventions: Other: Shoulder rehabilitation exercises and aerobic exercises

INTERVENTIONS:
Other: Shoulder rehabilitation exercises and aerobic exercises — SRG group: the group will only perform mobility and strengthening exercises involving the shoulder complex.
  ARG group: The ARG group will perform the shoulder rehabilitation protocol presented above combined with the aerobic exercise program that will last 20 minutes per session at 40% of the reserve heart rate (HRC), progressing up to 40 minutes with a maximum of 60% of the HRC in the last two weeks, according to the recommendations for patients with type 2 DM proposed in the American College of Sports Medicine Guidelines.

SUMMARY:
Goals: to compare the effects of two distinct rehabilitation protocols (conventional shoulder musculoskeletal rehabilitation combined with aerobic exercises versus solely conventional shoulder musculoskeletal rehabilitation) on shoulder pain, function, strength, kinematics and tendon thickness in patients with type 2 DM after 12 weeks of intervention and a subsequent follow up of 8 weeks. The secondary objective of this study will be to evaluate the association between AGEs accumulation and shoulder pain, function, strength, kinematics and tendon thickness in individuals with type 2 DM.

Methodology: is a single-blinded randomized controlled trial, in which all subjects with a clinical diagnosis of type 2 DM (with at least 1 year of diagnosis), of both sexes, between 40 and 70 years, presenting shoulder pain (uni or bilateral) for at least 3 months with a pain intensity score from 3 points on a numerical rating scale for pain intensity, will be invited to participate. The main outcomes of this study will include the AGEs accumulation through skin autofluorescence measurement; shoulder pain through NRS scales; shoulder function through SPADI questionnaire and range of motion measurement; isometric shoulder muscles strength through manual muscle dynamometer measurement; shoulder kinematics through three dimensional inertial units measurements; supraspinatus tendon thickness through ultrasound measurement. All these outcomes will be measured before and after the rehabilitation protocols. Participants will be randomly assigned to one of the two rehabilitation groups: specific shoulder rehabilitation protocol group (SRG); or 2) specific protocol of shoulder rehabilitation plus aerobic exercise group (ARG). All individuals will be evaluated before starting the rehabilitation protocol (baseline) and at the end of rehabilitation (post 12 weeks) and 8 weeks after the end of the rehabilitation (follow up). For the statistical analysis, to verify the effectiveness of protocols over time, a variance analysis (ANOVA) of mixed model with Bonferroni adjustment will be performed for pairwise comparisons. Variables that do not meet the ANOVA assumptions will be analyzed by the Mann-Whitney and Wilcoxon tests with Bonferroni correction a priori. In order to assess the secondary objective of the study, correlation tests depending on data distribution will be performed (Pearson or Spearman correlation tests). A simple linear regression analysis will also be performed in order to analyze how much the AGEs accumulation can explain the alterations in the musculoskeletal and biomechanical variables. The significance level will be set at 5%.

DETAILED DESCRIPTION:
SRG Protocol: shoulder rehabilitation protocol The protocol will be performed on a group with a maximum of 5 participants. Exercises intensity and difficulty will progress after completing 1 month of assistance, by increasing range of motion and loads (dumbbells) or resistance (elastic bands) in the exercises that are convenient. Each session will consist of 6 stages: 1) Pendulum exercise (10 repetitions - maintenance for 20 seconds); 2) Slide in flexion of the arms on the table (2 sets of 10 repetitions, maintenance in maximum range for 20 seconds); 3) Abduction and adduction (2 sets of 10 repetitions, maintenance for 20 seconds); 4) Wall slide - sliding of the arms on the wall (2 series of 10 repetitions, maintenance of 20 seconds); 5) Internal and external rotation (2 sets of 10 repetitions, maintenance for 20 seconds); 6) Elongation of the posterior capsule (cross-body) and pectoralis minor (3 repetitions of 30 seconds each). Pain will be evaluated during the protocol using the visual analog scale (VAS). The exercises proposed in this protocol are those that have already demonstrated in the literature an improvement in the function, strength, range of motion, and pain of the shoulder complex of the general population (27, 58).

The intensity and duration of the resistance exercises will be monitored by the physical therapist using heart rate monitors and adjusted to follow the same heart rate progression as outlined below for the aerobic group (ARG). In this manner, the average energy expenditure for both exercise groups will be similar. The protocol duration will be between 30-35 minutes. All sessions will be supervised by a physiotherapist with experience in physical exercise.

ARG group: Shoulder rehabilitation protocol combined to aerobic exercise program The ARG group will perform the shoulder rehabilitation protocol presented above combined with the aerobic exercise program. The aerobic program will last 20 minutes per session at 40% of the reserve heart rate (HRC), progressing up to 40 minutes with a maximum of 60% of the HRC in the last two weeks, according to the recommendations for patients with type 2 DM proposed in the American College of Sports Medicine Guidelines (59). The program will be carried out in groups of 4 participants and each session will consist of 3 stages: 1) Warm-up (5 min): patients will perform stretches of the main muscle groups; 2) Aerobic exercise in the treadmill with continuous heart rate monitors (Polar Electro Oy, Kempele, Finland), which will be used to adjust workload to achieve the target heart rate (15-40 min); 3) Cooldown (5 min): Stretching of the main muscle groups worked during the sessions and relaxation. In this way, the rehabilitation protocol of ARG group will last a total of approximately 90 minutes maximum. Before and after each session, blood pressure, heart rate and subjective perception of effort will be measured. During sessions, heart rate will be monitored by a heart rate monitor (Polar Vantage, Finland), and perceived exertion will be measured using the Borg CR20 scale, which should remain approximately between 11-13 (59). All sessions will be supervised by a physiotherapist with experience in physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be participants with a clinical diagnosis of type 2 DM (with at least 1 year of diagnosis), of both sexes, between 30 and 70 years, presenting shoulder pain (uni or bilateral) for at least 3 months with a pain intensity score from 3 points on a numerical rating scale for pain intensity (PI-NRS).

Exclusion Criteria:

* It will be excluded participants with a history of stabilization or surgical shoulder repair; recent history of fracture of the upper limb; cognitive deficits that make it difficult to understand verbal commands; who have undergone shoulder rehabilitation in the past 6 months; neuromuscular diseases; central nervous system diseases and rheumatological arthropathies.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
HbA1c - Glycated hemoglobin | 12-weeks
  HbA1c (mmol/mol) will be evaluated through blood tests that will be performed in the clinical laboratory of the University, at the beginning (before starting the treatment protocol), after the 12-week intervention (3-7 days after the last session) and after the 8-week follow-up.
lipid profile | 12-weeks
  lipid profile (mmol/L) will be evaluated through blood tests that will be performed in the clinical laboratory of the University, at the beginning (before starting the treatment protocol), after the 12-week intervention (3-7 days after the last session) and after the 8-week follow-up.
fasting glucose | 12-weeks
  fasting glucose (mmol/L) will be evaluated through blood tests that will be performed in the clinical laboratory of the University, at the beginning (before starting the treatment protocol), after the 12-week intervention (3-7 days after the last session) and after the 8-week follow-up.
AGEs accumulation measurement | 12-weeks
  Skin autofluorescence (nm wavelength) is considered as a substitute variable of AGEs accumulation. To perform this measurement, the AGE Reader (DiagnOptics, Groningen, the Netherlands) will be used, which non-invasively assesses skin autofluorescence.
Shoulder pain measurement | 12-weeks
  Shoulder pain will be evaluated through the numerical pain scale (Numerical Rating Scale 0 to 10, the higher the score, higher the pain).
Shoulder function measurement SPADI | 12-weeks
  The participant must respond to the SPADI questionnaire (Shoulder Pain and Disability Index - Spanish validated version).The SPADI score can range from 0 % indicating no pain or disability, to 100 % indicating severe pain and total disability
Shoulder function measurement Range of motion | 12-weeks
  the range of motion will be measured (in degrees) for all shoulder complex movements using a digital inclinometer (Acumar™, Lafayette Intrument Company, Lafayette, IN).
Isometric shoulder muscles strength measurement | 12-weeks
  Isometric muscle strength of the shoulder muscles will be assessed (in Newton) using a hand held dynamometer (HHD) (Lafayette Instrument, Lafayette, IN).
Shoulder three dimensional kinematics | 12-weeks
  Shoulder three-dimensional kinematics (in degrees) will be recorded (80 Hz) during arm elevation in the scapular plane and during a reaching over 90° functional task, using an inertial movement units system (IMU system) (MTW Awinda Xsens, Nexgen Ergonomics, Canada).
Supraspinatus tendon thickness measurement | 12-weeks
  Ultrasonographic measurement for each participant's supraspinatus tendon thickness (millimeters) will be scanned by using a Lumify Ultrasound in conjunction with a 4-12 MHz linear transducer (Philips Medical System).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Habechian FAP, Flores Quezada ME, Cools AM, Kjaer BH, Cuevas Cid RI, Zanca GG. Shoulder-specific rehabilitation combined with aerobic exercises versus solely shoulder-specific rehabilitation in patients with type 2 diabetes mellitus: study protocol for a randomized controlled superiority trial. Trials. 2022 Aug 17;23(1):678. doi: 10.1186/s13063-022-06647-5. PMID 35978380